CLINICAL TRIAL: NCT04873687
Title: Effectiveness of External Counter Pulsation (ECP) Therapy in Stable Angina Pectoris Patients; a Proof of Principal Clinical Trial
Brief Title: Effectiveness of ECP Therapy in Stable Angina Pectoris Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Principal Investigator, Badai Bhatara Tiksnadi, Head of Cardiovascular Prevention and Rehabilitation Clinic Dr. Hasan Sadikin General Hospital, Universitas Padjadjaran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Card-202103.01
Record Dates: First submitted 2021-04-24; First posted 2021-05-05 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Counterpulsation; Angina Pectoris
Keywords: External Counterpulsation; Stable Angina Pectoris; Indicated CABG; Global longitudinal strain; Ischemic response
MeSH Terms: conditions — Angina Pectoris; Angina, Stable | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: The intervention will be administered to eligible stable angina pectoris patients Dr. Hasan Sadikin General Hospital in a randomized manner neither of experiment or control group.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor and study statistician will not be aware of intervention assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm will comprise study participants who receive intervention therapy (i.e eligible stable angina pectoris patients in intervention arm who agree to participate)
  Interventions: Device: External Counter Pulsation (ECP) therapy
- Control (No Intervention): Eligible stable angina pectoris patients in the control arm will receive no intervention therapy

INTERVENTIONS:
Device: External Counter Pulsation (ECP) therapy — ECP therapy consist of 36 session, each session @1 hour/day, five days a week with initial pressure of 300mmHg
  Arms: Intervention

SUMMARY:
External Counterpulsation (ECP) is a non-invasive therapy using pressured cuff that is performed on patients with refractory stable angina pectoris to relieve symptoms and increase quality of life. In Indonesia, waiting time for getting coronary artery bypass grafting (CABG) procedure for revascularization treatment in stable angina pectoris patients is way longer than international recommendation which correlates with increase morbidity and mortality during the waiting time. Utilization of ECP for such patients who wait for CABG procedure is still unclear. The investigator aim to evaluate efficacy of addition of ECP compared with medical therapy alone for this population. The efficacy is evaluated using measurement from echocardiography result, treadmill test result, and clinical outcome. if applicable, examination of myocardial perfusion using nuclear examination will also be performed.

DETAILED DESCRIPTION:
Waiting time for elective CABG procedure in Indonesia is usually longer than six weeks, way longer than the European society of cardiology recommendation. During the waiting time, patients still complain of having troubling chest pain and at risk from 1.7% mortality even after optimal medical therapy. ECP is a non-invasive therapy using a pressured cuff performed on patients that have been utilized in refractory angina pectoris patients to relieve symptoms, increase the quality of life, and decrease future major adverse cardiac events (MACE).

This study is proof of principal clinical trial to evaluate the efficacy of addition ECP therapy after optimal medical therapy for stable angina pectoris patients waiting for CABG in Dr. Hasan Sadikin General Hospital, Bandung, Indonesia. Eligible patients will be informed about the study and randomized to the intervention arm. Patients in the experimental arm will undergo ECP therapy consisting of 36 sessions, each session @1 hour/day, five days a week with an initial pressure of 300mmHg. No intervention will be given to patients in the control arm.

The primary and secondary endpoint is the change in variables measured before and after the intervention is fully implemented. The primary endpoint variables are global longitudinal strain (GLS), Left ventricular ejection fraction (LVEF), Time to ST-Segment depression, duration of treadmill test, the Canadian cardiovascular society (CCS) score, and the Seattle angina questionnaire (SAQ) score. The secondary endpoint variable will be myocardial perfusion score measured as Summed Rest Score, Summed Stress Score, Summed Difference Score, Myocardial Micro-alternation Index (MMI), the level of Vascular Endothelial Growth Factor (VEGF), microRNA-92a (miR-92a), NT pro BNP, Troponin, incidence of MACE, general quality of life based on questionnaire The Indonesian EQ-5D-5L, and effectiveness of ECP for stable angina pectoris patients with pharmaco-economy studies. This change will then be compared between the intervention experimental arm and control arm.

Safety oversight by a Data and Safety Monitoring Board (DSMB) will be conducted by independent parties. Internal Data Monitoring Committee (DMC) will be established to oversee the study, focused on data quality. Quality control (QC) procedures will be implemented beginning with the data entry system. Data QC checks that will be run on the database will be automatically generated weekly, and any quality issues identified will be reviewed by the DMC a plan put in place for resolution.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Diagnosed with stable angina pectoris
* Anatomic vessel disease (VD) lesion with 2VD/3VD
* Indicated for CABG and in waiting list of CABG procedure; or refuse for CABG and choose medical therapy only; or patients who are decided by the responsible doctor for medical treatment alone because of the high risks of CABG surgery.
* Not planned to urgent CABG
* Minimum optimal medical therapy within 2 weeks
* Able and willing to sign informed consent and comply with study procedures
* The patient lives in Bandung City and its neighborhood
* Retired patient; or not actively working during working hours; or willing to take the time to participate in research.

Exclusion Criteria:

* Congestive Heart Failure
* Chronic heart failure with Functional Class NYHA III - IV
* LVEF <35%
* Unprotected left main stenosis >50%
* Blood pressure >180/110mmHg
* Acute coronary syndrome
* Acute Heart Failure
* Severe aorta regurgitation
* Malignant arrhythmia
* Atrial fibrillation
* Premature ventricular complex
* Peripheral occlusive artery disease
* Phlebitis
* Deep vein thrombosis
* Hemorrhagic diathesis
* Severe chronic kidney disease
* Aortic aneurysm
* Abdominal aneurysm
* Osteoarthritis
* Low back pain
* Pregnancy
* Registered as other clinical study participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Global Longitudinal Strain (GLS) | At baseline and week 7 (post intervention)
  GLS is a parameter captured through transthoracic echocardiography. GLS was calculated as the mean peak longitudinal systolic strain of all the LV segments, consistent with American Society of Echocardiography (ASE) guidelines.
Change in Left Ventricular Ejection Fraction (LVEF) | At baseline and week 7 (post intervention)
  LVEF is a parameter captured through transthoracic echocardiography. LVEF was calculated by Simpson biplane method
Change in Time to mm ST-segment Depression | At baseline and week 7 (post intervention)
  Time to induce significant ST-segment Depression using treadmill exercise test
Change in Duration of Treadmill Test | At baseline and week 7 (post intervention)
  Maximally tolerated time of treadmill exercise test using Bruce protocol or Modified Bruce protocol
Change in CCS score | At baseline and week 7 (post intervention)
  Degree of presenting chest pain symptoms using the Canadian cardiovascular society (CCS) class score. CCS class score ranging from 1 (mild) to 4 (severe)
Change in Seattle Angina Questionnaire (SAQ) Score | At baseline and week 7 (post intervention)
  Quality of life based on The Seattle Angina Questionnaire measurement. The possible range of scores for each of the five subscales is 0 to 100, with higher scores indicating better quality of life. A change of 10 points in any of the subscales is considered to be clinically important.

SECONDARY OUTCOMES:
Change in Summed Rest Score (SRS) | At baseline and week 7 (post intervention)
  Summed Rest Score is part of myocardial perfusion parameters of SPECT myocardial perfusion defects examination. The score are accumulated from 17 polar map segment. each segment scored. the extent and severity of perfusion deficits while rest ranging from 0 to 4 with higher score mean worse clinical apperance.
Change in Summed Stress Score (SSS) | At baseline and week 7 (post intervention)
  Summed Stress Score is part of myocardial perfusion parameters of SPECT myocardial perfusion defects examination. The score are accumulated from 17 polar map segment. each segment scored. the extent and severity of perfusion deficits while stress ranging from 0 to 4 with higher score mean worse clinical apperance.
Change in Summed Difference Score (SDS) | At baseline and week 7 (post intervention)
  Summed Difference Score is part of myocardial perfusion parameters of SPECT myocardial perfusion defects examination. SDS can be calculated by subtracting the SRS from the SSS (SDS = SSS - SRS). This measure is used to describe the degree to which the deficit/ischemia is reversible. An SDS score of 0-1 indicates no ischemia; 2-4 points indicate mild ischemia; 5-6 points indicate moderate ischemia; while 7 or more points indicate severe ischemia.
Myocardial Micro-alternation Index (MMI) | At baseline and week 7 (post intervention)
  Myocardial Micro-alternation Index is part of ECG dispersion mapping (ECG-DM)
The level of Vascular Endothelial Growth Factor (VEGF) | At baseline and week 7 (post intervention)
  Blood tests were carried out to determine levels of VEGF using ELISA and quantitative reverse transcription-polymerase chain reaction (qRT-PCR). The measurement unit is pg/ml.
The level of microRNA-92a (miR-92a) | At baseline and week 7 (post intervention)
  Blood tests were carried out to determine levels of miR-92a using ELISA and quantitative reverse transcription-polymerase chain reaction (qRT-PCR).
The level of NT pro BNP and Troponin | At baseline and week 7 (post intervention)
  Blood tests were carried out to determine levels of NT pro BNP (measurement unit pg/ml).
The level of Troponin | At baseline and week 7 (post intervention)
  Blood tests were carried out to determine levels of Troponin (measurement unit ng/ml).
Change in Quality of Life | At baseline and week 7 (post intervention)
  Quality of life based on Questionnaire The Indonesian EQ-5D-5L, is a questionnaire used to assess the quality of life of angina pectoris patients undergoing ECP treatment, allowing us to determine how much money can be saved in extending a patient's life for one year. It consists of five assessment domains, which are walking ability, self-care, usual activities, pain/discomfort, and anxiety/depression. The normal range is 0-1, with a score of 1 indicating the best quality of life.
Major Adverse Cardiac Event (MACE) | 2 years
  Number of incidence of Major adverse cardiac event
Effectiveness of ECP for stable angina pectoris patients | At baseline and week 7 (post intervention)
  Effectiveness of ECP for stable angina pectoris patients is based on pharmacoeconomics. The assessment will use the ICER formula, comparing optimal medication therapy from both healthcare and national insurance perspectives, taking into account about nominal outcomes, clinical outcomes, and patient quality of life outcomes. The results from the formula will then be input into a diagram to determine whether they fall into quadrant 1, 2, 3, or 4 (the best outcome is if it falls into quadrant 2).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad R Akbar, MD, FIHA., Principal Investigator — Universitas Padjadjaran
Locations (1):
- Dr. Hasan Sadikin General Hospital, Bandung, West Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arora RR, Chou TM, Jain D, Fleishman B, Crawford L, McKiernan T, Nesto RW. The multicenter study of enhanced external counterpulsation (MUST-EECP): effect of EECP on exercise-induced myocardial ischemia and anginal episodes. J Am Coll Cardiol. 1999 Jun;33(7):1833-40. doi: 10.1016/s0735-1097(99)00140-0. PMID 10362181
- [Background] Wu E, Desta L, Brostrom A, Martensson J. Effectiveness of Enhanced External Counterpulsation Treatment on Symptom Burden, Medication Profile, Physical Capacity, Cardiac Anxiety, and Health-Related Quality of Life in Patients With Refractory Angina Pectoris. J Cardiovasc Nurs. 2020 Jul/Aug;35(4):375-385. doi: 10.1097/JCN.0000000000000638. PMID 31929322
- [Background] Subramanian R, Nayar S, Meyyappan C, Ganesh N, Chandrakasu A, Nayar PG. Effect of Enhanced External Counter Pulsation Treatment on Aortic Blood Pressure, Arterial Stiffness and Ejection Fraction in Patients with Coronary Artery Disease. J Clin Diagn Res. 2016 Oct;10(10):OC30-OC34. doi: 10.7860/JCDR/2016/23122.8743. Epub 2016 Oct 1. PMID 27891374
- [Background] Zhang C, Liu X, Wang X, Wang Q, Zhang Y, Ge Z. Efficacy of Enhanced External Counterpulsation in Patients With Chronic Refractory Angina on Canadian Cardiovascular Society (CCS) Angina Class: An Updated Meta-Analysis. Medicine (Baltimore). 2015 Nov;94(47):e2002. doi: 10.1097/MD.0000000000002002. PMID 26632696
- [Background] Head SJ, da Costa BR, Beumer B, Stefanini GG, Alfonso F, Clemmensen PM, Collet JP, Cremer J, Falk V, Filippatos G, Hamm C, Kappetein AP, Kastrati A, Knuuti J, Kolh P, Landmesser U, Laufer G, Neumann FJ, Richter DJ, Schauerte P, Taggart DP, Torracca L, Valgimigli M, Wijns W, Witkowski A, Windecker S, Juni P, Sousa-Uva M. Adverse events while awaiting myocardial revascularization: a systematic review and meta-analysis. Eur J Cardiothorac Surg. 2017 Aug 1;52(2):206-217. doi: 10.1093/ejcts/ezx115. PMID 28472484
- [Background] Rampengan SH, Prihartono J, Siagian M, Immanuel S. The Effect of Enhanced External Counterpulsation Therapy and Improvement of Functional Capacity in Chronic Heart Failure patients: a Randomized Clinical Trial. Acta Med Indones. 2015 Oct;47(4):275-82. PMID 26932695